CLINICAL TRIAL: NCT00148343
Title: Functional Electrical Stimulation for Footdrop in Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, John Chae, MD, Prof, Chair Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB04-00104; R01HD044816 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Hemiplegia
Keywords: hemiplegia; hemiparesis; stroke; foot-drop; electrical stimulation; ankle-foot-orthosis
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- ODFS (Experimental): Odstock Dropped-Foot Stimulator (ODFS)
  Interventions: Device: Odstock Dropped-Foot Stimulator (ODFS); Procedure: Traditional Physical Therapy Treatment
- Standard of Care (inc. AFO) (Active Comparator): Conventional Standard of Care (which may include a study-specific Custom Molded Hinged Ankle Foot Orthosis (AFO)) [Traditional Physical Therapy Treatment]
  Interventions: Other: Conventional Standard of Care; Procedure: Traditional Physical Therapy Treatment

INTERVENTIONS:
Device: Odstock Dropped-Foot Stimulator (ODFS) — Device implementation & use for ~13 weeks (until 2nd Outcomes Assessment (1st post-treatment Outcomes Assessment)). The ODFS then will be returned to the investigators.
  Arms: ODFS
Other: Conventional Standard of Care — Conventional standard of care (which may include implementation & use of a study-specific Custom Molded Hinged Ankle Foot Orthosis (AFO)) for ~13 weeks (until 2nd Outcomes Assessment (1st post-treatment Outcomes Assessment)). The AFO, if implemented, may continue to be used afterwards since it is an element of the standard of care for this patient population.
  Arms: Standard of Care (inc. AFO)
Procedure: Traditional Physical Therapy Treatment — Traditional physical therapy treatment for 12 weeks.

SUMMARY:
The objective of this research is to determine if electrical stimulation can improve the strength and coordination of the lower limb muscles, and the walking ability of stroke survivors.

The knowledge gained from this study may lead to enhancements in the quality of life of stroke survivors by improving their neurological recovery and mobility. The results may lead to substantial changes in the standard of care for the treatment of lower limb hemiparesis after stroke.

DETAILED DESCRIPTION:
Hemiplegia is a major consequence of stroke and contributes significantly to the physical disability of stroke survivors. Foot-drop, or inability to dorsiflex the paretic ankle during the swing phase of gait, and ankle instability during stance phase, are important gait abnormalities that contribute to reduced mobility among stroke survivors. In the United States, the standard of care in addressing these deficits is the custom molded ankle-foot-orthosis (AFO). However, evolving data now demonstrate that active repetitive movement training is the principal substrate for facilitating motor relearning after stroke. Motor relearning is defined as the reacquisition of motor ability after central nervous system injury. Thus, while an AFO may assist stroke survivors to ambulate in the short-term, it is possible that it also inhibits recovery in the long-term. Previous studies have demonstrated that active repetitive movement exercises mediated by neuromuscular electrical stimulation (NMES) facilitate motor relearning among stroke survivors. In particular, studies have reported that some chronic stroke survivors treated with a peroneal nerve stimulator for foot-drop experience sufficient recovery that they no longer need the peroneal nerve stimulator or an AFO for community ambulation. However, there are no blinded randomized clinical trials that rigorously evaluate the motor relearning effects of ambulation training with peroneal nerve stimulators. Thus, the primary aim of this project is to assess the effects of transcutaneous peroneal nerve stimulation on lower limb motor relearning among chronic stroke survivors. The secondary aim is to assess the effects of transcutaneous peroneal nerve stimulation on lower limb mobility (disability) and overall quality of life. A single-blinded randomized clinical trial will be carried out to assess the effects of ambulation training with a peroneal nerve stimulator among chronic stroke survivors compared to ambulation training with conventional standard of care (which may include an AFO). Subjects will be treated for 12 weeks and followed for a total of another 6 months. This project will determine the effectiveness of peroneal nerve stimulation in facilitating motor relearning and improving the mobility and quality of life of stroke survivors. This proposed approach is expected to improve patient outcome and challenge the present clinical paradigm of prescribing AFOs for stroke survivors with foot-drop.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors >90 days from most recent clinical hemorrhagic or nonhemorrhagic stroke
* Age: 18-80 years
* Unilateral hemiparesis
* Medically stable
* Sufficient endurance & motor ability to ambulate at least 30 feet continuously with minimal assistance [requiring contact guard to no more than 25% physical help] or less without the use of an AFO
* Berg Balance Scale score of 24 or greater without any assistive devices
* Ankle dorsiflexion strength of no greater than 4/5 on the Medical Research Council (MRC) scale while standing
* Demonstrate foot-drop during ambulation such that gait instability [need for supervision, physical assistance or assistive device (cane, walker) to maintain balance or prevent falls] or inefficient gait patterns [gait pattern manifesting "dragging" or "catching" of the affected toes during swing phase of gait, or use of compensatory strategies such as circumducting the affected limb, vaulting with the unaffected limb or hiking the affected hip to clear the toes] are exhibited
* Ankle dorsiflexion to at least neutral while standing in response to NMES of the common peroneal nerve without painful hypersensitivity to the NMES
* If using an AFO, willing to terminate its use and comply with study requirements

Exclusion Criteria:

* Require an AFO to maintain knee stability (prevention of knee flexion collapse) during stance phase of gait
* Edema of the affected lower limb which interferes with the safe and effective use of a peroneal nerve stimulator
* Skin breakdown of the affected lower limb which interferes with the safe and effective use of a peroneal nerve stimulator
* Absent sensation of the affected lower limb
* History of potentially fatal cardiac arrhythmias, such as ventricular tachycardia, supraventricular tachycardia, and rapid ventricular response atrial fibrillation with hemodynamic instability
* Demand pacemakers or any other implanted electronic systems
* Pregnant women
* Uncontrolled seizure disorder
* Parkinson's Disease
* Spinal cord injury
* Traumatic brain injury with evidence of motor weakness
* Multiple sclerosis
* Fixed ankle plantar flexor contracture
* Peroneal nerve injury at the fibular head as the cause of foot-drop
* Uncompensated hemineglect
* Severely impaired cognition and communication
* Painful hypersensitivity to NMES of the common peroneal nerve
* Inadequate social support (potential unlikeliness to comply with treatment & follow-up)
* History of Botulinum toxin (Botox) injection to either of the lower extremities within the 3 month period preceding study entry
* Knee hyperextension (genu recurvatum) that cannot be adequately corrected with peroneal nerve stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-07; Primary Completion 2010-08-02 (Actual); Study Completion 2010-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Chae, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burridge JH, Taylor PN, Hagan SA, Wood DE, Swain ID. The effects of common peroneal stimulation on the effort and speed of walking: a randomized controlled trial with chronic hemiplegic patients. Clin Rehabil. 1997 Aug;11(3):201-10. doi: 10.1177/026921559701100303. PMID 9360032
- [Background] Burridge J, Taylor P, Hagan S, Swain I. Experience of clinical use of the Odstock dropped foot stimulator. Artif Organs. 1997 Mar;21(3):254-60. doi: 10.1111/j.1525-1594.1997.tb04662.x. PMID 9148719
- [Background] Burridge JH, McLellan DL. Relation between abnormal patterns of muscle activation and response to common peroneal nerve stimulation in hemiplegia. J Neurol Neurosurg Psychiatry. 2000 Sep;69(3):353-61. doi: 10.1136/jnnp.69.3.353. PMID 10945810
- [Background] Burridge JH, Wood DE, Taylor PN, McLellan DL. Indices to describe different muscle activation patterns, identified during treadmill walking, in people with spastic drop-foot. Med Eng Phys. 2001 Jul;23(6):427-34. doi: 10.1016/s1350-4533(01)00061-3. PMID 11551819
- [Background] Taylor PN, Burridge JH, Dunkerley AL, Wood DE, Norton JA, Singleton C, Swain ID. Clinical use of the Odstock dropped foot stimulator: its effect on the speed and effort of walking. Arch Phys Med Rehabil. 1999 Dec;80(12):1577-83. doi: 10.1016/s0003-9993(99)90333-7. PMID 10597809
- [Background] Taylor PN, Burridge JH, Dunkerley AL, Lamb A, Wood DE, Norton JA, Swain ID. Patients' perceptions of the Odstock Dropped Foot Stimulator (ODFS). Clin Rehabil. 1999 Oct;13(5):439-46. doi: 10.1191/026921599677086409. PMID 10498351
- [Background] Taylor P, Burridge J. Functional Electrical Stimulation - the Odstock Dropped Foot Stimulator. In: Sassoon R, ed. Understanding Stroke: Pardoe Blacker Publishing Ltd, 2002:72-78.
- [Background] Taylor P. The use of electrical stimulation for correction of dropped foot in subjects with upper motor neuron lesions. Advances in Clinical Neurosciences and Rehabilitation 2002; 2:16-18.
- [Background] Chae J, Bethoux F, Bohine T, Dobos L, Davis T, Friedl A. Neuromuscular stimulation for upper extremity motor and functional recovery in acute hemiplegia. Stroke. 1998 May;29(5):975-9. doi: 10.1161/01.str.29.5.975. PMID 9596245
- [Background] Francisco G, Chae J, Chawla H, Kirshblum S, Zorowitz R, Lewis G, Pang S. Electromyogram-triggered neuromuscular stimulation for improving the arm function of acute stroke survivors: a randomized pilot study. Arch Phys Med Rehabil. 1998 May;79(5):570-5. doi: 10.1016/s0003-9993(98)90074-0. PMID 9596400
- [Background] Mann GE, Wright PA, Swain ID. Training effects of electrical stimulation and the conventional ankle foot orthosis in the correction of drop foot following stroke., 1st Annual Conference of FESnet, 2002.
- [Background] Taylor P, Mann G, Swain I. Does prior use of an Ankle Foot Orthosis (AFO) effect the response to use of the Odstock Dropped Foot Stimulator?, Institute of Physics and Engineering in Medicine (IPEM) Annual Scientific Meeting, Bath, U.K., September 15-17, 2003:89-90.
- [Background] Buurke JH, Roetenberg D, Kleissen RFM, Hermens HJ. Early recovery of gait after stroke, 3rd World Congress in Neurological Rehabilitation, Venice, Italy, April 2-6, 2002, 2002.
- [Background] El-Hayek K, Quinn A, Berezovskiy R, Santing J, Harley M, Chae J. Relationship between lower limb motor impairment and ambulation function among chronic stroke survivors. Submitted.
- [Background] Teasell RW, Bhogal SK, Foley NC, Speechley MR. Gait retraining post stroke. Top Stroke Rehabil. 2003 Summer;10(2):34-65. doi: 10.1310/UDXE-MJFF-53V2-EAP0. PMID 13680517
- [Background] Teasell RW, Foley NC, Bhogal SK, Speechley MR. An evidence-based review of stroke rehabilitation. Top Stroke Rehabil. 2003 Spring;10(1):29-58. doi: 10.1310/8YNA-1YHK-YMHB-XTE1. PMID 12970830
- [Background] International Society for Prosthetics and Orthotics. Consensus Conference on
- [Background] LIBERSON WT, HOLMQUEST HJ, SCOT D, DOW M. Functional electrotherapy: stimulation of the peroneal nerve synchronized with the swing phase of the gait of hemiplegic patients. Arch Phys Med Rehabil. 1961 Feb;42:101-5. No abstract available. PMID 13761879
- [Background] Waters RL, McNeal D, Perry J. Experimental correction of footdrop by electrical stimulation of the peroneal nerve. J Bone Joint Surg Am. 1975 Dec;57(8):1047-54. PMID 1081538
- [Background] Waters RL, McNeal DR, Clifford B. Correction of footdrop in stroke patients via surgically implanted peroneal nerve stimulator. Acta Orthop Belg. 1984 Mar-Apr;50(2):285-95. No abstract available. PMID 6741512
- [Background] Kljajic M, Malezic M, Acimovic R, Vavken E, Stanic U, Pangrsic B, Rozman J. Gait evaluation in hemiparetic patients using subcutaneous peroneal electrical stimulation. Scand J Rehabil Med. 1992 Sep;24(3):121-6. PMID 1411357
- [Background] van der Aa HE, Bultstra G, Verloop AJ, Kenney L, Holsheimer J, Nene A, Hermens HJ, Zilvold G, Buschman HP. Application of a dual channel peroneal nerve stimulator in a patient with a "central" drop foot. Acta Neurochir Suppl. 2002;79:105-7. doi: 10.1007/978-3-7091-6105-0_23. PMID 11974972
- [Background] Merletti R, Andina A, Galante M, Furlan I. Clinical experience of electronic peroneal stimulators in 50 hemiparetic patients. Scand J Rehabil Med. 1979;11(3):111-21. PMID 315098
- [Background] Granat MH, Maxwell DJ, Ferguson AC, Lees KR, Barbenel JC. Peroneal stimulator; evaluation for the correction of spastic drop foot in hemiplegia. Arch Phys Med Rehabil. 1996 Jan;77(1):19-24. doi: 10.1016/s0003-9993(96)90214-2. PMID 8554468
- [Background] Takebe K, Kukulka C, Narayan MG, Milner M, Basmajian JV. Peroneal nerve stimulator in rehabilitation of hemiplegic patients. Arch Phys Med Rehabil. 1975 Jun;56(6):237-9. PMID 1079717
- [Background] Takebe K, Basmajian JV. Gait analysis in stroke patients to assess treatments of foot-drop. Arch Phys Med Rehabil. 1976 Jul;57(1):305-10. PMID 1084734
- [Background] Stefancic M, Rebersek M, Merletti R. The therapeutic effects of the Ljublijana functional electrical brace. Eur Medicophys 1976; 12:1-9.
- [Background] Carnstam B, Larsson LE, Prevec TS. Improvement of gait following functional electrical stimulation. I. Investigations on changes in voluntary strength and proprioceptive reflexes. Scand J Rehabil Med. 1977;9(1):7-13. PMID 302481
- [Background] Sullivan SB. Stroke. In: Sullivan SB, ed. Physical Rehabilitation: Assessment and Treatment. Philadelphia: F. A. Davis Company, 1994:327-360.
- [Background] Verbeke G, Molenbergh G. Linear mixed models for longitudinal data. New York: Springer-Verlag, 2000.
- [Background] Harrell FE. Regression modeling strategies. New York: Springer-Verlag, 2001.
- [Derived] Sheffler LR, Taylor PN, Bailey SN, Gunzler DD, Buurke JH, IJzerman MJ, Chae J. Surface peroneal nerve stimulation in lower limb hemiparesis: effect on quantitative gait parameters. Am J Phys Med Rehabil. 2015 May;94(5):341-57. doi: 10.1097/PHM.0000000000000269. PMID 25802966
- [Derived] Sheffler LR, Taylor PN, Gunzler DD, Buurke JH, Ijzerman MJ, Chae J. Randomized controlled trial of surface peroneal nerve stimulation for motor relearning in lower limb hemiparesis. Arch Phys Med Rehabil. 2013 Jun;94(6):1007-14. doi: 10.1016/j.apmr.2013.01.024. Epub 2013 Feb 8. PMID 23399456
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects screened over 5-yr study period: 469. Subjects completing informed consent and eligibility eval: 158. Subjects enrolled: 110. Last date of enrollment:10/27/2009. Final date subject study completion: 8/2/2010. All subject screening, enrollment, and study participation took place at an academic medical center.
Pre-assignment Details: Enrolled subjects (n=110) were stratified by presence or absence of dorsiflexion, based on clinical exam, prior to randomization into treatment and control groups. No enrolled subjects were excluded from the trial prior to assignment to groups.
Groups:
- Peroneal Nerve Stimulation (PNS): The peroneal nerve stimulator used in this study was the Odstock Dropped-Foot Stimulator (ODFS).
- Standard of Care (no Device or Ankle Foot Orthosis): Conventional Standard of Care was defined as either 1) no device or 2) a custom molded hinged ankle foot orthosis (AFO). Standard of care intervention device was determined based on clinical indication.
Period: Overall Study
Arm/Group | Peroneal Nerve Stimulation (PNS) | Standard of Care (no Device or Ankle Foot Orthosis)
Started | 54 | 56
Completed | 39 | 45
Not Completed | 15 | 11
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Physician Decision | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Peroneal Nerve Stimulation: Odstock Dropped Foot Stimulator
- Standard of Care: No device or ankle foot orthosis
- Total: Total of all reporting groups
Arm/Group | Peroneal Nerve Stimulation | Standard of Care | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 51 | 98
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (12.2) | 53.2 (10.1) | 53.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 30 | 37 | 67
Region of Enrollment [Number; unit: participants]
  United States | 54 | 56 | 110

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Motor Assessment (FMA)
Description: Lower limb motor impairment as measured by the lower limb portion of the Fugl-Meyer Assessment (FMA) which consists of 17 items, with a maximum possible score of 34 points, with lower scores indicating higher impairment. Each item was answered using a 3-point ordinal scale (0 = cannot perform, 1 = can partially perform, 2 = can fully perform).
Time Frame: Weeks 0, 12, 24, 36
Population: For intent-to-treat analysis, all participants who were randomized and completed baseline assessments were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peroneal Nerve Stimulation | Standard of Care
Number analyzed (Participants) | 53 | 55
units on a scale
  Baseline | 20.1 (5.9) | 20.3 (6.0)
  12- weeks | 21.5 (6.27) | 21.18 (5.72)
  24- weeks | 21.26 (6.05) | 21.17 (5.58)
  36 weeks | 21.93 (5.84) | 21.02 (5.69)
Statistical Analysis 1: Comparison: Peroneal Nerve Stimulation vs Standard of Care; Test type: Superiority or Other; Slope = 1.26, 95% CI 2-sided [-0.2 to 2.75], Standard Error of Mean 0.76 — Mixed model analysis. Slope is in reference to treatment x time interaction for full 36 weeks

2. Secondary Outcome: Steps Per Minute
Description: The number of steps taken by participants in one minute
Time Frame: Weeks 0, 12, 24, 36
Measure: Mean (Standard Deviation); unit: Steps/Min
Arm/Group | Peroneal Nerve Stimulation | Standard of Care
Number analyzed (Participants) | 54 | 56
Steps/Min
  Baseline | 65.0 (22) | 66.7 (22.7)
  12-weeks | 67.4 (21.5) | 72.6 (22.6)
  24-weeks | 69.3 (26.35) | 72.0 (23.16)
  36-weeks | 70.84 (26.83) | 73.74 (22.73)
Statistical Analysis 1: Comparison: Peroneal Nerve Stimulation vs Standard of Care; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = -5.07, 95% CI 2-sided [-10.05 to -0.09], Standard Error of Mean 2.54 — Slope is in reference to from baseline to end of follow-up at 36 weeks

3. Secondary Outcome: Modified Emory Functional Ambulation Profile(mEFAP)
Description: The mEFAP comprises 5 individually timed tasks performed over different environmental terrains. The subtasks include (1) a 5-meter walk on a hard floor; (2) a 5-meter walk on a carpeted surface; (3) rising from a chair, a 3-meter walk, and return to a seated position (the "timed up-and-go" test); (4) traversing a standardized obstacle course; and (5) ascending and descending 5 stairs. The mEFAP is performed with or without the use of an orthotic device or an AD. Manual assistance (MA) is provided as necessary. The subject can use rails when climbing the stairs. The 5 timed subscores are added to derive a total score in seconds.
Time Frame: Weeks 0, 12, 24, 36
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Peroneal Nerve Stimulation | Standard of Care
Number analyzed (Participants) | 54 | 56
seconds
  Baseline | 121.54 (86.59) | 118.39 (74.10)
  12- weeks | 107.92 (78.80) | 93.47 (73.02)
  24-weeks | 110.81 (81.89) | 97.25 (71.4)
  36-weeks | 111.81 (83.16) | 96.20 (65.20)
Statistical Analysis 1: Comparison: Peroneal Nerve Stimulation vs Standard of Care; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = 0.31, 95% CI 2-sided [-14.096 to 14.716], Standard Error of Mean 7.35 — Slope is in reference to start of treatment to end of follow up at 36 weeks

4. Secondary Outcome: Stroke-Specific Quality of Life Scale (SS-QOL)
Description: The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke. Patients must respond to each question of the SS-QOL with reference to the past week. It is a self-report scale containing 49 items in 12 domains: Mobility, Energy, Upper extremity function, Work/productivity, Mood, Self-care, Social roles, Family roles, Vision, Language, Thinking, Personality. There are 11 subscales.
  Items are rated on a 5-point Likert scale with higher scores indicate better functioning. The overall SS-QOL summary score (summation of all items) is presented here. Scores range from 49-245.
Time Frame: Weeks 0, 12, 24, 36
Measure: Mean (Standard Deviation); unit: Summary Score
Arm/Group | Peroneal Nerve Stimulation | Standard of Care
Number analyzed (Participants) | 54 | 56
Summary Score
  Baseline | 179.12 (35.73) | 175.30 (40.67)
  12-weeks | 191.62 (42.39) | 185.42 (34.76)
  24-weeks | 195.66 (38.25) | 184.87 (38.88)
  36-weeks | 190.23 (44.73) | 182.95 (39.76)
Statistical Analysis 1: Comparison: Peroneal Nerve Stimulation vs Standard of Care; Test type: Superiority; Slope = -1.95, 95% CI 2-sided [-12.79 to 8.89], Standard Error of Mean 5.53 — Mixed models analysis. Slope refers to baseline to final follow up at 36 weeks

5. Secondary Outcome: Gait Speed
Time Frame: baseline, 12, 24 and 36 weeks
Measure: Mean (Standard Deviation); unit: meters/sec
Arm/Group | Peroneal Nerve Stimulation | Standard of Care
Number analyzed (Participants) | 54 | 56
meters/sec
  Baseline | 0.35 (0.20) | 0.40 (0.24)
  12-weeks | 0.40 (0.25) | 0.47 (0.24)
  24-weeks | 0.44 (0.28) | 0.46 (0.25)
  36-weeks | 0.44 (0.28) | 0.47 (0.24)
Statistical Analysis 1: Comparison: Peroneal Nerve Stimulation vs Standard of Care; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = 0.006, 95% CI 2-sided [-0.045 to 0.057], Standard Error of Mean 0.026 — Slope is in reference to baseline to end of follow-up at 36 weeks

ADVERSE EVENTS:
Arm/Group | Peroneal Nerve Stimulation | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 21/54 | 7/56
Other Adverse Events (participants affected / at risk) | 39/54 | 20/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peroneal Nerve Stimulation (N=54) | Standard of Care (N=56)
infection (Infections and infestations) | 0 (0) | 1 (1)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Fall (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (2)
Neurologic change (Nervous system disorders) | 7 (8) | 0 (0)
Cardiac (Cardiac disorders) | 4 (4) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 0 (0) | 1 (1)
Urologic (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peroneal Nerve Stimulation (N=54) | Standard of Care (N=56)
Fall (Injury, poisoning and procedural complications) | 25 (38) | 15 (24)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 13 (16) | 4 (4)
Neurologic (Nervous system disorders) | 2 (3) | 3 (3)
Skin (Skin and subcutaneous tissue disorders) | 17 (21) | 4 (9)

LIMITATIONS AND CAVEATS:
1. Uneven randomization with respect to dorsiflexion status and mEFAP at baseline.
2. High drop out rate of 30% for the ODFS and 20% for usual care
3. Optimal dose and duration of treatment unknown
4. Activity monitor on ODFS and AFO not reliable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No